CLINICAL TRIAL: NCT00665366
Title: A 12-Week, Multicenter, Randomized, Double-Blind, Placebo-Controlled Study To Evaluate the Efficacy and Safety of Adjunctive Aripiprazole Therapy in the Treatment of Mania in Bipolar I Disorder Patients Treated on Valproate or Lithium and in Need of Further Clinical Improvement
Brief Title: Study to Evaluate the Efficacy and Safety of Aripiprazole Administered With Lithium or Valproate Over 12 Weeks in the Treatment of Mania in Bipolar I Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Collaborators: Otsuka America Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CN138-502; EudraCT number 2007-005959-42
Record Dates: First submitted 2008-04-18; First posted 2008-04-23 (Estimated); Results first posted 2013-02-04 (Estimated); Last update posted 2013-12-02 (Estimated); Status verified 2013-02

CONDITIONS: Bipolar Disorder Mania
MeSH Terms: interventions — Aripiprazole; Lithium; Valproic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo + valproate or lithium (Placebo Comparator): Participants randomly received placebo (1:1 to study drug) as adjunctive therapy to current ongoing treatment with valproate or lithium for 12 weeks.
  Interventions: Drug: Placebo; Drug: Lithium; Drug: Valproate
- Aripiprazole + valproate or lithium (Active Comparator): Participants randomly received aripiprazole as adjunctive therapy to current ongoing treatment with valproate or lithium for 12 weeks. Aripiprazole was provided in 5-, 10-, or 15-mg oral tablets and administered at a starting dose of 5 mg per day for Week 1. For Weeks 2 through 3, the dose was titrated up to 10 mg per day, and for Weeks 4 through 6, the dose increased to 15 mg per day. Flexible doses of either 15 or 30 mg per day were administered for Weeks 7 through 12. If participants were unable to tolerate the dose of 15 mg per day of study drug, the dose was decreased to 10 mg per day for Weeks 7 through 12.
  Interventions: Drug: Aripiprazole; Drug: Lithium; Drug: Valproate

INTERVENTIONS:
Drug: Aripiprazole — 5-, 10-, or 15-mg oral tablets in titrated doses for 12 weeks
  Other Names: Abilify; BMS-337039
  Arms: Aripiprazole + valproate or lithium
Drug: Placebo — Tablets, Oral, 0 mg, once daily, 12 weeks
  Arms: Placebo + valproate or lithium
Drug: Lithium — Participant's ongoing dose
Drug: Valproate — Participant's ongoing dose

SUMMARY:
The purpose of the study is to determine whether aripiprazole provides additional clinical benefit to patients with Bipolar I disorder when combined with lithium or valproate over 12 weeks.

ELIGIBILITY:
Key inclusion criteria:

* Clinical diagnosis of bipolar I disorder mania, manic or mixed episode, with or without psychotic features
* Current ongoing lithium or valproate treatment with the possibility of benefiting, based on the investigator's clinical judgment, from adjunctive treatment with aripiprazole
* Therapeutic serum levels of lithium or valproate and a Young Mania Rating Total Score of 16 or higher at screening and baseline
* Participants taking current lithium or valproate treatment combined with antipsychotic medication other than aripiprazole are acceptable, provided that the other antipsychotic medication is washed out at least 3 days prior to the blood draw for therapeutic plasma levels of lithium and valproate determination. Long-acting antipsychotics must be washed out prior to entering the double-blind treatment.

Key exclusion criteria:

* Women of childbearing potential who are unwilling or unable to use an acceptable method to avoid pregnancy for the entire study period and for up to 4 weeks after the last dose of investigational product
* A diagnosis of delirium, dementia, amnesia or other cognitive disorder, or a psychotic disorder
* Current diagnosis of delirium, dementia, a cognitive disorder (ie, amnesia), or a psychotic disorder (ie, schizophrenia or schizoaffective disorder)
* Current diagnosis of bipolar II disorder, bipolar disorder not otherwise specified, or any other primary psychiatric disorder other than bipolar I disorder mania
* Thyroid pathology
* Demonstrated cocaine abuse or dependence within the past 3 months prior to screening.
* History of neuroleptic malignant syndrome from antipsychotic agents
* Manic symptoms that investigator considers refractory to treatment
* Previous nonresponsive (by investigator judgment) to aripiprazole for manic symptoms
* Significant risk of suicide based on history, mental status exam, or investigator judgment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 493 (Actual)
Dates: Start 2008-06; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (65):
- Austria (2):
  - Local Institution, Salzburg
  - Local Institution, Vienna
- Czechia (3):
  - Local Institution, Hradec Králové
  - Local Institution, Litoměřice
  - Local Institution, Prague
- France (15):
  - Local Institution, Beaupuy
  - Local Institution, Brumath
  - Local Institution, Château-Gontier
  - Local Institution, Clermont-Ferrand
  - Local Institution, Dijon
  - Local Institution, Dole
  - Local Institution, Jonzac
  - Local Institution, Le Vésinet
  - Local Institution, Montpellier
  - Local Institution, Nîmes
  - Local Institution, Paris
  - Local Institution, Reims
  - Local Institution, Saint-Nazaire
  - Local Institution, Sotteville-lès-Rouen
  - Local Institution, Strasbourg
- Germany (2):
  - Local Institution, Ellwangen
  - Local Institution, Ostfildern
- Greece (4):
  - Local Institution, Athens
  - Local Institution, Leros
  - Local Institution, Nea Ionia-Athens
  - Local Institution, Tripoli
- Hungary (3):
  - Local Institution, Budapest
  - Local Institution, Győr
  - Local Institution, Gyula
- Italy (10):
  - Local Institution, Campobasso
  - Local Institution, Foggia
  - Local Institution, Foligno (Pg)
  - Local Institution, Genova
  - Local Institution, La Spezia
  - Local Institution, Milan
  - Local Institution, Napoli
  - Local Institution, Pisa
  - Local Institution, Roma
  - Local Institution, Sant'Arsenio (Salerno)
- Poland (5):
  - Local Institution, Choroszcz
  - Local Institution, Gdansk
  - Local Institution, Krakow
  - Local Institution, Poznan
  - Local Institution, Swiecie N/Wisla
- Romania (3):
  - Local Institution, Bucharest
  - Local Institution, Cluj-Nappoca
  - Local Institution, Iași
- Russia (7):
  - Local Institution, Khot'kovo
  - Local Institution, Krasnodar
  - Local Institution, Moscow
  - Local Institution, Rostov-on-Don
  - Local Institution, Saint Petersburg
  - Local Institution, Samara
  - Local Institution, Tomsk
- South Africa (5):
  - Local Institution, Johannesburg, Gauteng
  - Local Institution, Soweto, Gauteng
  - Local Institution, Vereeniging, Gauteng
  - Local Institution, Pinetown, KwaZulu-Natal
  - Local Institution, Cape Town, Western Cape
- Spain (3):
  - Local Institution, Barcelona
  - Local Institution, Madrid
  - Local Institution, Murcia
- Turkey (Türkiye) (3):
  - Local Institution, Ankara
  - Local Institution, Antalya
  - Local Institution, Denizli

REFERENCES:
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 493 participants enrolled, 370 were randomized, and 369 received treatment with double-blind study medication.
Period: Overall Study
Arm/Group | Placebo + Valproate or Lithium | Aripiprazole + Valproate or Lithium
Started | 189 (Participants randomized) | 181 (Participants randomized)
Completed | 131 | 122
Not Completed | 58 | 59
Not completed — Lack of Efficacy | 11 | 10
Not completed — Adverse Event | 25 | 23
Not completed — Withdrawal by Subject | 11 | 14
Not completed — Lost to Follow-up | 3 | 5
Not completed — Poor compliance/noncompliance | 3 | 5
Not completed — Pregnancy | 1 | 0
Not completed — No longer meets study criteria | 0 | 1
Not completed — Other reasons | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo + Valproate or Lithium | Aripiprazole + Valproate or Lithium | Total
Number analyzed (Participants) | 189 | 181 | 370
Age Continuous [Mean (Standard Deviation); unit: Years] | 44.92 (12.99) | 44.37 (12.13) | 44.65 (12.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 99 | 101 | 200
  Male | 90 | 80 | 170
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 179 | 172 | 351
  Black/African American | 6 | 6 | 12
  Asian | 1 | 2 | 3
  Other | 3 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Total Score on the Young Mania Rating Scale (YMRS) (LOCF Data Set)
Description: The YMRS is a clinician-administered scale, consisting of 11 multiple choice items, and used to assess a patient's manic symptoms and clinical condition over the previous 48 hours. Total scores range from 0 to 60, with 12 or greater signifying hypomania or mania. Each item is given a severity rating ranging from 0 to 8 or 0 to 4. Items for the scale are based on the core symptoms of mania: elevated mood, increased motor activity, sexual interest, sleep, irritability, speech (rate and amount), language-though disorder, content, disruptive-aggressive behavior, appearance, and insight. Scores for each item reflect the severity of that symptom in the patient. The test is administered during a clinical interview typically lasting 15-30 minutes. LOCF=last observation carried forward.
Time Frame: Baseline to Week 12
Population: All randomized participants who received at least 1 dose of study medication and who had at least 1 efficacy evaluation after the start of study drug.
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo + Valproate or Lithium | Aripiprazole + Valproate or Lithium
Number analyzed (Participants) | 186 | 176
Units on a scale | -11.54 (0.78) | -13.57 (0.78)
Statistical Analysis 1: Comparison: Placebo + Valproate or Lithium vs Aripiprazole + Valproate or Lithium; Test type: Superiority or Other; p = 0.058, ANCOVA; Mean Difference (Final Values) = -2.04, 95% CI 2-sided [-4.14 to 0.07]

2. Secondary Outcome: Change From Baseline in Score on Clinical Global Impression-Bipolar Version (CGI-BP) Severity of Illness (Mania) Scale (LOCF Data Set)
Description: Adjusted mean change. The CGI-BP is a scale used to assess a clinician's impression of a patient's illness. Each patient is rated at baseline and at subsequent visits on items related to severity of depression, mania, and overall bipolar illness. The CGI-BP is a 7-point scale, with scores ranging from 1=normal/not ill to 7=very severely ill. Higher total score indicates greater severity of illness. LOCF=last observation carried forward.
Time Frame: Baseline to Weeks 3, 6, 9, and 12
Population: All randomized participants who received at least 1 dose of study medication and who had at least 1 efficacy evaluation after the start of study drug. n=number of evaluable participants.
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo + Valproate or Lithium | Aripiprazole + Valproate or Lithium
Number analyzed (Participants) | 186 | 176
Units on a scale
  Week 3 (n=183, 174) | -0.97 (0.08) | -0.93 (0.08)
  Week 6 (n=186, 176) | -1.35 (0.09) | -1.46 (0.10)
  Week 9 (n=186, 176) | -1.55 (0.10) | -1.83 (0.11)
  Week 12 (n=186, 176) | -1.78 (0.11) | -2.07 (0.11)
Statistical Analysis 1: Comparison: Placebo + Valproate or Lithium vs Aripiprazole + Valproate or Lithium; Test type: Superiority or Other; p = 0.669, ANOVA/ANCOVA; Mean Difference (Net) = 0.05, 95% CI 2-sided [-0.16 to 0.25] — Week 3
Statistical Analysis 2: Comparison: Placebo + Valproate or Lithium vs Aripiprazole + Valproate or Lithium; Test type: Superiority or Other; p = 0.436, ANOVA/ANCOVA; Mean Difference (Net) = -0.10, 95% CI 2-sided [-0.36 to 0.16] — Week 6
Statistical Analysis 3: Comparison: Placebo + Valproate or Lithium vs Aripiprazole + Valproate or Lithium; Test type: Superiority or Other; p = 0.053, ANOVA/ANCOVA; Mean Difference (Net) = -0.28, 95% CI 2-sided [-0.56 to 0.00] — Week 9
Statistical Analysis 4: Comparison: Placebo + Valproate or Lithium vs Aripiprazole + Valproate or Lithium; Test type: Superiority or Other; p = 0.044, ANOVA/ANCOVA; Mean Difference (Final Values) = -0.30, 95% CI 2-sided [-0.59 to -0.01] — Week 12

3. Secondary Outcome: Change From Baseline in Score on Clinical Global Impression-Bipolar Version (CGI-BP) Severity of Illness (Depression) Scale (LOCF Data Set)
Description: as for outcome 2
Time Frame: Baseline to Weeks 3, 6, 9, and 12
Population: as for outcome 2
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo + Valproate or Lithium | Aripiprazole + Valproate or Lithium
Number analyzed (Participants) | 186 | 176
Units on a scale
  Week 3 (n=183, 174) | -0.01 (0.05) | -0.09 (0.05)
  Week 6 (n=186, 176) | -0.02 (0.06) | -0.01 (0.06)
  Week 9 (n=186, 176) | -0.04 (0.07) | 0.11 (0.07)
  Week 12 (n=186, 176) | -0.03 (0.08) | 0.14 (0.08)
Statistical Analysis 1: Comparison: Placebo + Valproate or Lithium vs Aripiprazole + Valproate or Lithium; Test type: Superiority or Other; p = 0.240, ANOVA/ANCOVA model; Mean Difference (Net) = -0.08, 95% CI 2-sided [-0.22 to 0.06] — Week 3
Statistical Analysis 2: Comparison: Placebo + Valproate or Lithium vs Aripiprazole + Valproate or Lithium; Test type: Superiority or Other; p = 0.843, ANOVA/ANCOVA model; Mean Difference (Net) = 0.02, 95% CI 2-sided [-0.15 to 0.19] — Week 6
Statistical Analysis 3: Comparison: Placebo + Valproate or Lithium vs Aripiprazole + Valproate or Lithium; Test type: Superiority or Other; p = 0.117, ANOVA/ANCOVA model; Mean Difference (Net) = 0.16, 95% CI 2-sided [-0.04 to 0.35] — Week 9
Statistical Analysis 4: Comparison: Placebo + Valproate or Lithium vs Aripiprazole + Valproate or Lithium; Test type: Superiority or Other; p = 0.109, ANOVA/ANCOVA model; Week 12; Median Difference (Final Values) = 0.17, 95% CI 2-sided [-0.04 to 0.38]

4. Secondary Outcome: Change From Baseline in Score on Clinical Global Impression-Bipolar Version (CGI-BP) Severity of Illness (Overall) Scale at Week 12 (LOCF Data Set)
Description: Adjusted mean change. The CGI-BP is scale used to assess a clinician's impression of a patient's illness. Each patient is rated at baseline and at subsequent visits on items related to severity of depression, mania, and overall bipolar illness. The CGI-BP is a 7-point scale, with scores ranging from 1=normal/not ill to 7=very severely ill. Higher total score indicates greater severity of illness. LOCF=last observation carried forward.
Time Frame: Baseline to Week 12
Population: as for outcome 2
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo + Valproate or Lithium | Aripiprazole + Valproate or Lithium
Number analyzed (Participants) | 186 | 176
Units on a scale | -1.51 (0.11) | -1.59 (0.11)
Statistical Analysis 1: Comparison: Placebo + Valproate or Lithium vs Aripiprazole + Valproate or Lithium; Test type: Superiority or Other; p = 0.567, ANOVA/ANCOVA model; Week 12; Mean Difference (Final Values) = -0.08, 95% CI 2-sided [-0.37 to 0.20]

5. Secondary Outcome: Change From Baseline in Total and Subscale Scores on the Functional Assessment Short Test (FAST)(LOCF Data Set)
Description: The FAST is an interview-administered instrument used to assess the main functioning problems that patients with bipolar disorder experience. Participants are rated at Baseline, Week 3, Week 6, Week 9, and Week 12/End of Study Visit. The FAST consists of 24 items that assess impairment or disability in 6 specific areas of functioning, categorized as the subscales: autonomy, occupational functioning, cognitive functioning, financial issues, interpersonal (IP) relationships, and leisure time. All items are rated using a 4-point scale, 0=no difficulty, 1=mild difficulty, 2=moderate difficulty, and 3=severe difficulty. The global score is the sum of the scores of all items and ranges from 0 (0*24)to 96 (4*24). The higher the global score, the higher the level of impairment. function=functioning. LOCF=last observation carried forward.
Time Frame: Baseline to Weeks 3, 6, 9, and 12
Population: All randomized participants who received at least 1 dose of study medication and who had at least 1 outcomes research evaluation after the start of study drug. n=number of evaluable participants.
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo + Valproate or Lithium | Aripiprazole + Valproate or Lithium
Number analyzed (Participants) | 189 | 181
Units on a scale
  Total score: Week 3 (n=179, 169) | -5.68 (0.86) | -5.00 (0.87)
  Total score: Week 6 (n=182, 171) | -8.59 (0.98) | -6.93 (0.99)
  Total score: Week 9 (n=182, 171) | -9.18 (1.06) | -7.71 (1.07)
  Total score: Week 12 (n=182, 171) | -10.39 (1.09) | -8.51 (1.10)
  Autonomy score: Week 3 (n=179, 169) | -0.93 (0.18) | -0.93 (0.18)
  Autonomy score: Week 6 (n=182, 171) | -1.44 (0.19) | -1.11 (0.19)
  Autonomy score: Week 9 (n=182, 171) | -1.56 (0.21) | -1.20 (0.21)
  Autonomy score: Week 12 (n=182, 171) | -1.84 (0.21) | -1.45 (0.21)
  Occupational function score: Week 3 (n=179, 169) | -0.65 (0.25) | -1.00 (0.25)
  Occupational function score: Week 6 (n=182, 171) | -1.23 (0.29) | -1.40 (0.29)
  Occupational function score: Week 9 (n=182, 171) | -1.20 (0.30) | -1.22 (0.30)
  Occupational function score: Week 12 (n=182, 171) | -1.49 (0.30) | -1.24 (0.30)
  Cognitive function score: Week 3 (n=179, 169) | -1.33 (0.23) | -0.99 (0.23)
  Cognitive function score: Week 6 (n=182, 171) | -2.12 (0.26) | -1.46 (0.26)
  Cognitive function score: Week 9 (n=182, 171) | -2.30 (0.26) | -1.68 (0.27)
  Cognitive function score: Week 12 (n=182, 171) | -2.59 (0.27) | -1.91 (0.28)
  IP relationships score: Week 3 (n=179,169) | -1.57 (0.25) | -1.33 (0.26)
  IP relationships score: Week 6 (n=182, 171) | -2.20 (0.28) | -1.91 (0.29)
  IP relationships score: Week 9 (n=182, 171) | -2.41 (0.31) | -2.14 (0.31)
  IP relationships score: Week 12 (n=182, 171) | -2.57 (0.31) | -2.31 (0.31)
  Leisure time score: Week 3 (n=179, 169) | -0.50 (0.11) | -0.28 (0.11)
  Leisure time score: Week 6 (n=182, 171) | -0.53 (0.13) | -0.34 (0.13)
  Leisure time score: Week 9 (n=182, 171) | -0.52 (0.13) | -0.52 (0.13)
  Leisure time score: Week 12 (n=182, 171) | -0.68 (0.13) | -0.59 (0.13)
  Financial issues score: Week 3 (n=179, 169) | -0.78 (0.12) | -0.48 (0.12)
  Financial issues score: Week 6 (n=182, 171) | -1.16 (0.12) | -0.76 (0.13)
  Financial issues score: Week 9 (n=182, 171) | -1.25 (0.13) | -0.99 (0.13)
  Financial issues score: Week 12 (n=182, 171) | -1.30 (0.12) | -1.07 (0.13)
Statistical Analysis 1: Comparison: Placebo + Valproate or Lithium vs Aripiprazole + Valproate or Lithium; Test type: Superiority or Other; p = 0.566, ANCOVA; Mean Difference (Final Values) = 0.68, 95% CI 2-sided [-1.66 to 3.03] — Total score: Week 3
Statistical Analysis 2: Comparison: Placebo + Valproate or Lithium vs Aripiprazole + Valproate or Lithium; Test type: Superiority or Other; p = 0.221, ANCOVA; Mean Difference (Final Values) = 1.66, 95% CI [-1.00 to 4.32] — Total score: Week 6
Statistical Analysis 3: Comparison: Placebo + Valproate or Lithium vs Aripiprazole + Valproate or Lithium; Test type: Superiority or Other; p = 0.315, ANCOVA; Mean Difference (Final Values) = 1.47, 95% CI 2-sided [-1.40 to 4.35] — Total score: Week 9
Statistical Analysis 4: Comparison: Placebo + Valproate or Lithium vs Aripiprazole + Valproate or Lithium; Test type: Superiority or Other; p = 0.212, ANCOVA; Mean Difference (Final Values) = 1.88, 95% CI 2-sided [-1.08 to 4.84] — Total score: Week 12
Statistical Analysis 5: Comparison: Placebo + Valproate or Lithium vs Aripiprazole + Valproate or Lithium; Test type: Superiority or Other; p = 0.991, ANCOVA; Mean Difference (Final Values) = 0.00, 95% CI 2-sided [-0.49 to 0.48] — Autonomy score: Week 3
Statistical Analysis 6: Comparison: Placebo + Valproate or Lithium vs Aripiprazole + Valproate or Lithium; Test type: Superiority or Other; p = 0.201, ANCOVA; Mean Difference (Final Values) = 0.34, 95% CI 2-sided [-0.18 to 0.85] — Autonomy score: Week 6
Statistical Analysis 7: Comparison: Placebo + Valproate or Lithium vs Aripiprazole + Valproate or Lithium; Test type: Superiority or Other; p = 0.198, ANCOVA; Mean Difference (Final Values) = 0.37, 95% CI 2-sided [-0.19 to 0.93] — Autonomy score: Week 9
Statistical Analysis 8: Comparison: Placebo + Valproate or Lithium vs Aripiprazole + Valproate or Lithium; Test type: Superiority or Other; p = 0.178, ANCOVA; Mean Difference (Final Values) = 0.39, 95% CI 2-sided [-0.18 to 0.96] — Autonomy score: Week 12
Statistical Analysis 9: Comparison: Placebo + Valproate or Lithium vs Aripiprazole + Valproate or Lithium; Test type: Superiority or Other; p = 0.311, ANCOVA; Mean Difference (Final Values) = -0.34, 95% CI 2-sided [-1.01 to 0.32] — Occupational functioning score: Week 3
Statistical Analysis 10: Comparison: Placebo + Valproate or Lithium vs Aripiprazole + Valproate or Lithium; Test type: Superiority or Other; p = 0.671, ANCOVA; Mean Difference (Final Values) = -0.17, 95% CI 2-sided [-0.94 to 0.61] — Occupational functioning score: Week 6
Statistical Analysis 11: Comparison: Placebo + Valproate or Lithium vs Aripiprazole + Valproate or Lithium; Test type: Superiority or Other; p = 0.968, ANCOVA; Mean Difference (Final Values) = -0.02, 95% CI 2-sided [-0.83 to 0.79] — Occupational functioning score: Week 9
Statistical Analysis 12: Comparison: Placebo + Valproate or Lithium vs Aripiprazole + Valproate or Lithium; Test type: Superiority or Other; p = 0.546, ANCOVA; Mean Difference (Final Values) = 0.25, 95% CI 2-sided [-0.56 to 1.07] — Occupational functioning score: Week 12
Statistical Analysis 13: Comparison: Placebo + Valproate or Lithium vs Aripiprazole + Valproate or Lithium; Test type: Superiority or Other; p = 0.284, ANCOVA; Mean Difference (Final Values) = 0.34, 95% CI 2-sided [-0.28 to 0.96] — Cognitive functioning score: Week 3
Statistical Analysis 14: Comparison: Placebo + Valproate or Lithium vs Aripiprazole + Valproate or Lithium; Test type: Superiority or Other; p = 0.063, ANCOVA; Mean Difference (Final Values) = 0.66, 95% CI 2-sided [-0.04 to 1.35] — Cognitive functioning score: Week 6
Statistical Analysis 15: Comparison: Placebo + Valproate or Lithium vs Aripiprazole + Valproate or Lithium; Test type: Superiority or Other; p = 0.090, ANCOVA; Mean Difference (Final Values) = 0.62, 95% CI 2-sided [-0.10 to 1.34] — Cognitive functioning score: Week 9
Statistical Analysis 16: Comparison: Placebo + Valproate or Lithium vs Aripiprazole + Valproate or Lithium; Test type: Superiority or Other; p = 0.072, ANCOVA; Mean Difference (Final Values) = 0.68, 95% CI 2-sided [-0.06 to 1.42] — Cognitive functioning score: Week 12
Statistical Analysis 17: Comparison: Placebo + Valproate or Lithium vs Aripiprazole + Valproate or Lithium; Test type: Superiority or Other; p = 0.499, ANCOVA; Mean Difference (Final Values) = 0.24, 95% CI 2-sided [-0.45 to 0.93] — Interpersonal relationships score: Week 3
Statistical Analysis 18: Comparison: Placebo + Valproate or Lithium vs Aripiprazole + Valproate or Lithium; Test type: Superiority or Other; p = 0.457, ANCOVA; Mean Difference (Final Values) = 0.29, 95% CI 2-sided [-0.48 to 1.06] — Interpersonal relationships score: Week 6
Statistical Analysis 19: Comparison: Placebo + Valproate or Lithium vs Aripiprazole + Valproate or Lithium; Test type: Superiority or Other; p = 0.525, ANCOVA; Mean Difference (Final Values) = 0.27, 95% CI [-0.56 to 1.10] — Interpersonal relationships score: Week 9
Statistical Analysis 20: Comparison: Placebo + Valproate or Lithium vs Aripiprazole + Valproate or Lithium; Test type: Superiority or Other; p = 0.544, ANCOVA; Mean Difference (Final Values) = 0.26, 95% CI 2-sided [-0.58 to 1.09] — Interpersonal relationships score: Week 12
Statistical Analysis 21: Comparison: Placebo + Valproate or Lithium vs Aripiprazole + Valproate or Lithium; Test type: Superiority or Other; p = 0.149, ANCOVA; Mean Difference (Final Values) = 0.22, 95% CI 2-sided [-0.08 to 0.52] — Leisure time score: Week 3
Statistical Analysis 22: Comparison: Placebo + Valproate or Lithium vs Aripiprazole + Valproate or Lithium; Test type: Superiority or Other; p = 0.264, ANCOVA; Mean Difference (Final Values) = 0.19, 95% CI 2-sided [-0.15 to 0.54] — Leisure time score: Week 6
Statistical Analysis 23: Comparison: Placebo + Valproate or Lithium vs Aripiprazole + Valproate or Lithium; Test type: Superiority or Other; p = 0.988, ANCOVA; Mean Difference (Final Values) = 0.00, 95% CI 2-sided [-0.35 to 0.35] — Leisure time score: Week 9
Statistical Analysis 24: Comparison: Placebo + Valproate or Lithium vs Aripiprazole + Valproate or Lithium; Test type: Superiority or Other; p = 0.641, ANCOVA; Mean Difference (Final Values) = 0.08, 95% CI 2-sided [-0.27 to 0.44] — Leisure time score: Week 12
Statistical Analysis 25: Comparison: Placebo + Valproate or Lithium vs Aripiprazole + Valproate or Lithium; Test type: Superiority or Other; p = 0.068, ANCOVA; Mean Difference (Final Values) = 0.29, 95% CI 2-sided [-0.02 to 0.61] — Financial issues score: Week 3
Statistical Analysis 26: Comparison: Placebo + Valproate or Lithium vs Aripiprazole + Valproate or Lithium; Test type: Superiority or Other; p = 0.019, ANCOVA; Mean Difference (Final Values) = 0.40, 95% CI 2-sided [0.07 to 0.74] — Financial issues score: Week 6
Statistical Analysis 27: Comparison: Placebo + Valproate or Lithium vs Aripiprazole + Valproate or Lithium; Test type: Superiority or Other; p = 0.136, ANCOVA; Mean Difference (Final Values) = 0.26, 95% CI 2-sided [-0.08 to 0.60] — Financial issues score: Week 9
Statistical Analysis 28: Comparison: Placebo + Valproate or Lithium vs Aripiprazole + Valproate or Lithium; Test type: Superiority or Other; p = 0.18, ANCOVA; Mean Difference (Final Values) = 0.23, 95% CI [-0.11 to 0.57] — Financial issues score: Week 12

6. Secondary Outcome: Percentage of Participants Showing A Response From Baseline on the Young Mania Rating Scale (YMRS)(OC Data Set)
Description: Response on the YMRS is defined as a 50% or greater improvement from baseline in YMRS total score. The YMRS is clinician-administered and consists of 11 multiple choice items. It is used to assess a patient's manic symptoms and clinical condition over the previous 48 hours. Total scores range from 0 to 60, with 12 or greater signifying hypomania or mania. Each item is given a severity rating ranging from 0 to 8 or 0 to 4. Items for the scale are based on the core symptoms of mania: elevated mood, increased motor activity, sexual interest, sleep, irritability, speech (rate and amount), language-thought disorder, content, disruptive-aggressive behavior, appearance, and insight. Scores for each item reflect the severity of that symptom in the patient. The test is administered during a clinical interview typically lasting 15-30 minutes. OC=observed cases.
Time Frame: Baseline to Weeks 3, 6, 9, and 12
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo + Valproate or Lithium | Aripiprazole + Valproate or Lithium
Number analyzed (Participants) | 186 | 176
Percentage of participants
  Week 3 (n=183, 174) | 26.2 | 29.3
  Week 6 (n=186, 176) | 46.2 | 49.4
  Week 9 (n=186, 176) | 53.8 | 64.2
  Week 12 (n=186, 176) | 61.3 | 68.8
Statistical Analysis 1: Comparison: Placebo + Valproate or Lithium vs Aripiprazole + Valproate or Lithium; Test type: Superiority or Other; p = 0.466, Ration of response; Risk Ratio (RR) = 1.13, 95% CI 2-sided [0.81 to 1.59] — Week 3
Statistical Analysis 2: Comparison: Placebo + Valproate or Lithium vs Aripiprazole + Valproate or Lithium; Test type: Superiority or Other; p = 0.540, Risk ratio; Risk Ratio (RR) = 1.07, 95% CI 2-sided [0.86 to 1.32] — Week 6
Statistical Analysis 3: Comparison: Placebo + Valproate or Lithium vs Aripiprazole + Valproate or Lithium; Test type: Superiority or Other; p = 0.060, Risk ratio; Risk Ratio (RR) = 1.17, 95% CI 2-sided [0.99 to 1.38] — Week 9
Statistical Analysis 4: Comparison: Placebo + Valproate or Lithium vs Aripiprazole + Valproate or Lithium; Test type: Superiority or Other; p = 0.289, Risk ratio; Risk Ratio (RR) = 1.07, 95% CI 2-sided [0.94 to 1.23]

7. Secondary Outcome: Percentage of Participants Showing Remission in the Young Mania Rating Scale (YMRS) Score From Baseline (LOCF Data Set)
Description: Remission is defined as a YMRS total score of 12 or less. The YMRS is clinician-administered and consists of 11 multiple choice items. It is used to assess a patient's manic symptoms and clinical condition over the previous 48 hours. Total scores range from 0 to 60, with 12 or greater signifying hypomania or mania. Each item is given a severity rating ranging from 0 to 8 or 0 to 4. Items for the scale are based on the core symptoms of mania: elevated mood, increased motor activity, sexual interest, sleep, irritability, speech (rate and amount), language-thought disorder, disruptive-aggressive behavior, appearance, and insight. Scores for each item reflect the severity of that symptom in the patient. The test is administered during a clinical interview typically lasting 15-30 minutes. LOCF=last observation carried forward.
Time Frame: Baseline to Weeks 3,6, 9, and 12
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo + Valproate or Lithium | Aripiprazole + Valproate or Lithium
Number analyzed (Participants) | 186 | 176
Percentage of participants
  Week 3 (n=183, 174) | 30.6 | 31.0
  Week 6 (n=186, 176) | 48.9 | 51.7
  Week 9 (n=186, 176) | 57.0 | 65.9
  Week 12 (n=186, 176) | 64.0 | 69.9
Statistical Analysis 1: Comparison: Placebo + Valproate or Lithium vs Aripiprazole + Valproate or Lithium; Test type: Superiority or Other; p = 0.909, Risk ratio (RR); Risk Ratio (RR) = 1.02, 95% CI 2-sided [0.75 to 1.39] — Week 3
Statistical Analysis 2: Comparison: Placebo + Valproate or Lithium vs Aripiprazole + Valproate or Lithium; Test type: Superiority or Other; p = 0.573, RR; Risk Ratio (RR) = 1.06, 95% CI 2-sided [0.86 to 1.30] — Week 6
Statistical Analysis 3: Comparison: Placebo + Valproate or Lithium vs Aripiprazole + Valproate or Lithium; Test type: Superiority or Other; p = 0.080, RR; Risk Ratio (RR) = 1.16, 95% CI 2-sided [0.98 to 1.36] — Week 9
Statistical Analysis 4: Comparison: Placebo + Valproate or Lithium vs Aripiprazole + Valproate or Lithium; Test type: Superiority or Other; p = 0.211, RR; Risk Ratio (RR) = 1.10, 95% CI 2-sided [0.95 to 1.27] — Week 12

8. Secondary Outcome: Change From Baseline in Total Score on the Longitudinal Interval Follow-up Evaluation-Rating Impaired Functioning Tool (LIFE-RIFT)(OC Data Set and Week 12 LOCF Data Set)
Description: Adjusted mean change. The LIFE-RIFT total score ranges from 4 to 20 and is the sum of scores of 4 items: work, interpersonal relations, satisfaction, and recreation. A negative change score signifies improvement. OC=observed cases; LOCF=last observation carried forward.
Time Frame: Baseline to Weeks 6 and 12
Population: All randomized participants who received at least 1 dose of study medication and had at least 1 outcome research evaluation after the start of study drug. n=number of evaluable participants.
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo + Valproate or Lithium | Aripiprazole + Valproate or Lithium
Number analyzed (Participants) | 186 | 176
Units on a scale
  Week 6 (n=146, 135) | -2.13 (0.22) | -1.45 (0.23)
  Week 12 (n=123, 115) | -3.20 (0.28) | -2.37 (0.28)
  Week 12 (LOCF) (n=165, 150) | -2.30 (0.27) | -1.69 (0.28)
Statistical Analysis 1: Comparison: Placebo + Valproate or Lithium vs Aripiprazole + Valproate or Lithium; Test type: Superiority or Other; ANOVA/ANCOVA model; Mean Difference (Net) = 0.68, 95% CI 2-sided [0.07 to 1.29] — Week 6
Statistical Analysis 2: Comparison: Placebo + Valproate or Lithium vs Aripiprazole + Valproate or Lithium; Test type: Superiority or Other; p = 0.031, ANOVA/ANCOVA model; Mean Difference (Final Values) = 0.83, 95% CI 2-sided [0.08 to 1.58] — Week 12
Statistical Analysis 3: Comparison: Placebo + Valproate or Lithium vs Aripiprazole + Valproate or Lithium; Test type: Superiority or Other; p = 0.104, ANOVA/ANCOVA model; Mean Difference (Final Values) = 0.61, 95% CI 2-sided [-0.13 to 1.34] — Week 12 (LOCF)

9. Secondary Outcome: Participant Scores on Patient Global Impression Improvement (PGI-I) Scale (OC Data Set)
Description: Adjusted Mean Scores. The PGI-I is a self-administered 7-point scale, with scores ranging from 1 (very much improved) to 7 (very much worse), that assesses the improvement or worsening of a patient's illness relative to baseline at the beginning of the intervention. Scores: 1=very much improved; 2=much improved; 3=minimally improved; 4=no change; 5=minimally worse; 6=much worse; or 7=very much worse. OC=observed cases.
Time Frame: Baseline to Weeks 3, 6, 9, and 12
Population: as for outcome 5
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo + Valproate or Lithium | Aripiprazole + Valproate or Lithium
Number analyzed (Participants) | 186 | 176
Units on a scale
  Week 3 (n=178, 168) | 2.94 (0.10) | 2.99 (0.10)
  Week 6 (n=151, 140) | 2.39 (0.11) | 2.64 (0.11)
  Week 12 (n=127, 119) | 2.02 (0.12) | 2.24 (0.12)
  Week 12 (LOCF) (n=181, 173) | 2.60 (0.13) | 2.88 (0.13)
Statistical Analysis 1: Comparison: Placebo + Valproate or Lithium vs Aripiprazole + Valproate or Lithium; Test type: Superiority or Other; ANCOVA; Mean Difference (Net) = 0.06, 95% CI 2-sided [-0.21 to 0.32] — Week 3
Statistical Analysis 2: Comparison: Placebo + Valproate or Lithium vs Aripiprazole + Valproate or Lithium; Test type: Superiority or Other; ANCOVA; Mean Difference (Net) = 0.24, 95% CI 2-sided [-0.05 to 0.53] — Week 6
Statistical Analysis 3: Comparison: Placebo + Valproate or Lithium vs Aripiprazole + Valproate or Lithium; Test type: Superiority or Other; p = 0.197, ANCOVA; Mean Difference (Final Values) = 0.21, 95% CI 2-sided [-0.11 to 0.54] — Week 12
Statistical Analysis 4: Comparison: Placebo + Valproate or Lithium vs Aripiprazole + Valproate or Lithium; Test type: Superiority or Other; p = 0.111, ANCOVA; Mean Difference (Final Values) = 0.28, 95% CI 2-sided [-0.07 to 0.63] — Week 12 (LOCF)

10. Secondary Outcome: Change From Baseline in Participant Weight (OC Data Set and Week 12 LOCF Data Set)
Description: Adjusted mean change.OC=observed cases; LOCF=last observation carried forward.
Time Frame: Baseline to Weeks 3, 6, 9, and 12
Population: All randomized participants who received at least 1 dose of study medication. n=number of evaluable participants.
Measure: Mean (Standard Error); unit: Kilograms
Arm/Group | Placebo + Valproate or Lithium | Aripiprazole + Valproate or Lithium
Number analyzed (Participants) | 186 | 176
Kilograms
  Week 3 (n=177, 171) | -0.06 (0.16) | 0.14 (0.15)
  Week 6 (n=152,144) | -0.02 (0.20) | 0.29 (0.21)
  Week 9 (n=142, 128) | 0.07 (0.26) | -0.01 (0.26)
  Week 12 (n=133, 123) | 0.22 (0.29) | 0.02 (0.29)
  Week 12 (LOCF) (n=183, 174) | 0.11 (0.24) | 0.11 (0.23)
Statistical Analysis 1: Comparison: Placebo + Valproate or Lithium vs Aripiprazole + Valproate or Lithium; Test type: Superiority or Other; p = 0.983, ANOVA/ANCOVA model; Mean Difference (Final Values) = 0.01, 95% CI 2-sided [-0.63 to 0.64] — Week 12 LOCF

11. Secondary Outcome: Percentage of Participants With Relevant Weight Gain or Weight Loss From Baseline at Week 12 (LOCF Data Set)
Description: Relevant weight gain=7% or greater increase in weight; relevant weight loss=7% or greater decrease in weight. LOCF=last observation carried forward.
Time Frame: Baseline to Weeks 3, 6, 9, and12
Population: All randomized participants who received at least 1 dose of study medication. n=number of evaluable participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo + Valproate or Lithium | Aripiprazole + Valproate or Lithium
Number analyzed (Participants) | 186 | 176
Percentage of participants
  Weight gain: Week 12 (n=184,174) | 4.3 | 5.2
  Weight loss: Week 12 (n=184,174) | 2.7 | 4.0
Statistical Analysis 1: Comparison: Placebo + Valproate or Lithium vs Aripiprazole + Valproate or Lithium; Test type: Superiority or Other; Risk Ratio; Weight gain; Risk Ratio (RR) = 1.45, 95% CI 2-sided [0.57 to 3.71]

12. Secondary Outcome: Change From Baseline to Week 12 in Body Mass Index (BMI) (LOCF Data Set)
Description: BMI=Weight in kilograms /(Height in meters^2). LOCF=last observation carried forward.
Time Frame: Baseline to Week 12
Population: All randomized participants who received at least 1 dose of study medication. n=number of evaluable participants.
Measure: Median (Full Range); unit: kg/m^2
Arm/Group | Placebo + Valproate or Lithium | Aripiprazole + Valproate or Lithium
Number analyzed (Participants) | 186 | 176
kg/m^2 | 0.0 [0.0 to 0.3] | 0.0 [0.0 to 0.4]
Statistical Analysis 1: Comparison: Placebo + Valproate or Lithium vs Aripiprazole + Valproate or Lithium; Test type: Superiority or Other; p = 0.582, ANCOVA; Median Difference (Final Values) = 0.0

ADVERSE EVENTS:
Arm/Group | Aripiprazole | Placebo
Serious Adverse Events (participants affected / at risk) | 11/180 | 17/189
Other Adverse Events (participants affected / at risk) | 45/180 | 29/189
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Aripiprazole (N=180) | Placebo (N=189)
Hyperthermia (General disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 1
Coma (Nervous system disorders) | 1 | 0
Depression (Psychiatric disorders) | 4 | 2
Psychotic disorder (Psychiatric disorders) | 1 | 0
Alcohol abuse (Psychiatric disorders) | 0 | 2
Dysgeusia (Nervous system disorders) | 0 | 1
Grand mal convulsion (Nervous system disorders) | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 0 | 1
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 1
Vertebrobasilar insufficiency (Nervous system disorders) | 1 | 0
Bipolar I disorder (Psychiatric disorders) | 1 | 0
Mania (Psychiatric disorders) | 2 | 7
Rhinitis (Infections and infestations) | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Depression suicidal (Psychiatric disorders) | 1 | 0
Hand fracture (Injury, poisoning and procedural complications) | 0 | 1
Hypertension (Vascular disorders) | 0 | 1
Intentional drug misuse (Psychiatric disorders) | 0 | 1
Renal colic (Renal and urinary disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Suicidal ideation (Psychiatric disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Aripiprazole (N=180) | Placebo (N=189)
Insomnia (Psychiatric disorders) | 10 | 10
Depression (Psychiatric disorders) | 14 | 5
Nausea (Gastrointestinal disorders) | 10 | 5
Akathisia (Nervous system disorders) | 20 | 4
Headache (Nervous system disorders) | 5 | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.